CLINICAL TRIAL: NCT04447729
Title: A Multicenter, Open-label Pilot Study of the Efficacy and Safety of Fremanezumab for Treatment of Female Patients With Interstitial Cystitis-Bladder Pain Syndrome
Brief Title: A Study to Test if Fremanezumab Reduces Pain in Patients With Interstitial Cystitis-Bladder Pain Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to logistic reasons
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TV48125-CNS-20022
Record Dates: First submitted 2020-06-10; First posted 2020-06-25 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Interstitial Cystitis
Keywords: Interstitial cystitis-bladder pain syndrome (IC-BPS)
MeSH Terms: conditions — Cystitis, Interstitial | interventions — fremanezumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- fremanezumab (Experimental): Two doses, each dose consists of 4 injections with prefilled syringes
  Interventions: Drug: fremanezumab

INTERVENTIONS:
Drug: fremanezumab — Two doses, each dose consists of 4 injections with prefilled syringes

SUMMARY:
The primary objective of the study is to evaluate the efficacy of fremanezumab in reducing pain in patients with interstitial cystitis-bladder pain syndrome (IC-BPS).

A secondary efficacy objective of the study is to evaluate the effect of fremanezumab on other efficacy measures, including pain, voiding frequency, urinary symptoms, and quality of life.

And another secondary objective of the study is to evaluate the safety and tolerability of fremanezumab administered subcutaneously in adult patients with IC-BPS.

The planned active study period is 8 weeks; the entire planned study duration for each patient is 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* has a diagnosis of IC-BPS according to the American Urological Association endorsed criteria for a duration of ≥6 months to ≤15 years
* has IC-BPS with moderate to severe bladder pain and urinary frequency
* has urinary frequency of ≥8 voids/day
* has had a cystoscopy within 6months before screening with report indicating absence of Hunner lesion(s). A patient who has not had a cystoscopy within 6months may undergo cystoscopy, at the physician's discretion, and be rescreened for study entry.
* has persistent symptoms despite an adequate trial of 3 months of dietary counseling and modification
* has a body mass index within 18.5 to 39 kg/m2 and a body weight ≥99 lbs.
* has non-pharmacologic interventions (such as physical therapy, pelvic floor massage, acupuncture, naturopathy, new initiation of mindfulness exercises, or cognitive behavioral therapy) that are unchanged for a minimum of 30 days before the screening visit
* if of childbearing potential, must meet any of the following criteria:

  * Patients must use 1 form of highly effective contraception with their partners during the entire study period and for 5 months after the last dose of the IMP
  * Sexual abstinence is only considered a highly effective method if defined as refraining from heterosexual intercourse in the defined period. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient. Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a study, and withdrawal are not acceptable methods of contraception.
  * Patients of childbearing potential must have a negative serum beta-human chorionic gonadotropin (β-HCG) pregnancy test at the screening visit (confirmed by urine dipstick β-HCG pregnancy test at baseline)

NOTE- Additional criteria apply; please contact the investigator for more information

Exclusion Criteria:

* has any of the following confounding conditions: bladder stones, lower ureteric stones, vaginal candidiasis for which treatment was completed less than 30 days before the screening visit, urethral diverticulum, incomplete bladder emptying, overactive bladder (ie, urinary urgency associated with urinary incontinence or fear of incontinence), radiation cystitis, tuberculosis cystitis, vaginitis, neurogenic bladder, or any other condition/disease which, in the opinion of the investigator, could compromise subject safety or confound the collection or interpretation of study results
* is receiving any of the following treatments:

  * intravesical therapy of any kind, corticosteroid therapy, cyclosporine, or anti-tumor necrosis factor-α inhibitors within 2 months before the screening visit (visit 1)
  * cyclophosphamide or ketamine at any time
  * mAbs targeting the CGRP pathway (including erenumab, eptinezumab, galcanezumab, or fremanezumab) at any time; if the subject has participated in a clinical study with any of these mAbs, it has to be confirmed that the subject received placebo in order to be eligible for this study
* has a known history of previous urinary diversion procedure with or without bladder removal or bladder augmentation
* has a known history of a cystoscopy with bladder biopsy, hydrodistention, or fulguration or triamcinolone injection ≤3 months before the screening visit
* was diagnosed with and/or treated for chronic migraine, defined as headaches occurring on ≥15 days/28-day period at any time over the past 3 months
* is receiving prophylactic treatment for migraine disorders
* has a known history of hypersensitivity reactions to injected proteins, including mAbs and animal venoms, or a history of Stevens-Johnson syndrome/toxic epidermal necrolysis syndrome
* has a lifetime known history of any psychotic and/or bipolar disorder

NOTE- Additional criteria apply; please contact the investigator for more information

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2022-02-10 (Estimated); Study Completion 2022-02-10 (Estimated)

PRIMARY OUTCOMES:
change from baseline in weekly average of the daily worst pain scores over the past 24 hours as measured on the PI-NRS | Baseline to weeks 4 and 8
  Pain Intensity-Numerical Rating Scale (PI-NRS) - An 11-point scale that measures pain from 0 to 10 (0=no pain; 10=worst possible pain)

SECONDARY OUTCOMES:
change from baseline in the weekly average of the daily average pain PI-NRS score | Baseline, Week 4, and 8
  The Pain Intensity-Numerical Rating Scale (PI-NRS) is an 11-point scale that measures pain from 0 to 10 (0=no pain; 10=worst possible pain)
Change from baselines in frequency of voids over the past 24 hours and change in average void volume. | Baseline, Week 4, and 8
Patient's Global Impression of Change (PGIC) | Week 4 and 8
  Improvement is recorded on a 7-point scale, with 1 indicating very much improved, 4 indicating no change, and 7 indicating very much worse
change from baseline in the BPIC-SS assessed over the most recent past 7 days | Baseline, Week 4, and 8
  Bladder Pain/Interstitial Cystitis Symptom Score (BPIC-SS) an 8-item questionnaire. Scores may range from 0 to 38 (0=no symptoms, 38=most severe symptoms)
change from baseline in the (GUPI) Questionnaire assessed over the most recent past 7 days | Baseline, Week 4, and 8
  Genitourinary Pain Index (GUPI) Questionnaire. The GUPI has 10 pain items (total pain subscale score 0 to 23), 2 urinary symptom items (total urinary subscale score 0 to 10), and 3 QOL items (total QOL subscale score: 0 to 12).
percent of patients who do not complete treatment due to all causes | 8 weeks
number of adverse events during the study | 8 Weeks
Incidence of abnormal clinical laboratory test results (serum chemistry) | Baseline - Week 8
Incidence of abnormal hematology laboratory test results | Baseline - Week 8
Incidence of abnormal coagulation laboratory test results. | Baseline - Week 8
Incidence of abnormal urinalysis laboratory test results. | Baseline - Week 8
Incidence of abnormal vital signs | Baseline - Week 8
clinically significant changes in physical examination | Baseline - Week 8
  including body weight
Incidence of abnormal standard 12-lead electrocardiogram (ECG) findings | Baseline - Week 8
local tolerability at the injection site | Week 1 and Week 4
  Injection sites will be assessed for erythema, induration, ecchymosis, and pain immediately (ie, within 20 minutes ±5 minutes) and 1 hour (±15 minutes) after IMP administration.
number of hypersensitivity/anaphylaxis reactions | Baseline - Week 8
percent of patients who do not complete the treatment due to adverse events | Baseline - Week 8
anxiety and depression as measured by the HADS | Baseline - Week 8
  Hospital Anxiety and Depression Scale (HADS): Scale for both anxiety and depression scored separately: 8-10 Mild, 11-14 Moderate, 15-21 Severe
suicidal ideation and behavior as measured by the C-SSRS | Baseline - Week 8
  The Columbia-Suicide Severity Rating Scale (C-SSRS) captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Questions included the presence of the following: a wish to be dead; nonspecific active suicidal thoughts; actual suicide attempt; non-suicidal self-injurious behavior; interrupted attempt; aborted attempt; suicidal behavior; preparatory suicidal acts or behavior; and completed suicide.
  The most severe type of ideation (i.e., 1-5 with 1 being the least severe and 5 being the most severe.

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be reviewed for scientific merit, product approval status, and conflicts of interest. Patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.